CLINICAL TRIAL: NCT00254501
Title: Empowering Patients to Better Manage Diabetes Through Self-Care
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Oregon State University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Principal Investigator, Dale F Kraemer, Associate Professor, University of Florida
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OSU_COP_PP_0105; IRB Application 2979
Record Dates: First submitted 2005-11-14; First posted 2005-11-16 (Estimated); Results first posted 2016-07-22 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Type I or Type II Diabetes (Excludes Gestational Diabetes)
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care plus out-of-pocket cost waiver (Active Comparator): Patients received educational materials (handouts) in the mail. This was assumed to be of minimal effectiveness. Patients also received waiver of out-of-pocket expenses for diabetes care.
  Interventions: Behavioral: Educational materials
- EMPOWER (Experimental): Patients were scheduled for free counseling with pharmacists including medication, diet, and other self-management items. Patients also received waiver of out-of-pocket expenses for diabetes care.
  Interventions: Behavioral: Pharmacist Counseling

INTERVENTIONS:
Behavioral: Pharmacist Counseling — Patients were scheduled for free counseling with pharmacists including medication, diet, and other self-management items. Patients also received waiver of out-of-pocket expenses for diabetes care.
  Arms: EMPOWER
Behavioral: Educational materials — Patients received educational materials (handouts) in the mail. This was assumed to be of minimal effectiveness. Patients also received waiver of out-of-pocket expenses for diabetes care.
  Arms: Usual Care plus out-of-pocket cost waiver

SUMMARY:
This study will look at the impact of health insurance benefits on self management of diabetes for people with this condition. Studies have shown that when people with diabetes manage their disease better, they stay healthier. Our goal in this study is to help those with diabetes better manage their disease (self-care). We will compare two types of health insurance benefits in this study. We want to see if one set of benefits improves self-care more than the other one.

DETAILED DESCRIPTION:
The objective of this particular study is to determine if the addition of regular pharmacist visits to usual care can improve clinical outcomes in patients with diabetes. The central hypothesis is that a program overseen by community pharmacists that empowers patients to self-manage their diabetes will lead to improved clinical and humanistic outcomes and will be cost-effective. Strong preliminary data collected from other sites suggests that patient empowerment programs are effective at reducing hemoglobin A1C after 12 months and in reducing the total cost of care. This hypothesis will be tested by pursuing three specific aims to evaluate the impact of a pharmacist-administered diabetes patient empowerment program on:

1. clinical markers for diabetes and related metabolic disorders;
2. the cost of care and resource utilization; and
3. patient knowledge and perceived ability to manage diabetes. There is an additional specific aim to assess the pharmacists with respect to satisfaction with the training program and the overall project, the activities conducted in patient sessions, and the time taken to complete the visits in this study.

ELIGIBILITY:
Inclusion Criteria:

* diabetes (Type I or Type II)
* enrolled in health plan with participating employer
* age 18 or older
* willing and able to provide informed consent

Exclusion Criteria:

* gestational diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2005-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dale F Kraemer, Ph.D., Principal Investigator — Oregon State University, College of Pharmacy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kraemer DF, Kradjan WA, Bianco TM, Low JA. A randomized study to assess the impact of pharmacist counseling of employer-based health plan beneficiaries with diabetes: the EMPOWER study. J Pharm Pract. 2012 Apr;25(2):169-79. doi: 10.1177/0897190011418513. Epub 2011 Oct 10. PMID 21987530

RESULTS

PARTICIPANT FLOW:
Groups:
- Usual Care Plus Out-of-pocket Cost Waiver: Employees received a waiver of out-of-pocket expenses (copayments or co-insurance) for specified diabetes-related medications (including hypertensive and dyslipidemic medications) and physician visits. They also received printed educational materials at enrollment and about 3 months into the study.
- EMPOWER Group: Employees received the same waiver of out-of-pocket expenses and also received up to 12 monthly visits with a pharmacist for consulting on monitoring and other educational aspects of diabetes self-management.
Period: Overall Study
Arm/Group | Usual Care Plus Out-of-pocket Cost Waiver | EMPOWER Group
Started | 32 | 37
Completed | 31 | 36
Not Completed | 1 | 1
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Plus Out-of-pocket Cost Waiver | EMPOWER Group | Total
Number analyzed (Participants) | 31 | 36 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (9.2) | 55.6 (6.8) | 54.2 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 14 | 33
  Male | 12 | 22 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 31 | 34 | 65
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 1 | 1
  White | 30 | 32 | 62
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Education categories [Number; unit: participants]
  High school graduate | 5 | 4 | 9
  Some college | 17 | 15 | 32
  College graduate | 8 | 11 | 19
  At least a masters degree | 0 | 3 | 3
  Unspecified | 1 | 3 | 4
Income categories [Number; unit: participants]
  $15 000 to <$30 000 | 3 | 3 | 6
  $30 000 to <$50 000 | 11 | 12 | 23
  $50 000 to <$100 000 | 11 | 10 | 21
  $100 000 or more | 2 | 10 | 12
  Unspecified | 4 | 1 | 5
Hypertension [Number; unit: participants]
  Yes | 16 | 26 | 42
  No | 15 | 10 | 25
Dyslipidemia [Number; unit: participants]
  Yes | 16 | 25 | 41
  No | 15 | 11 | 26
Depression [Number; unit: participants]
  Yes | 10 | 6 | 16
  No | 21 | 30 | 51
On glucose-lowering therapy [Number; unit: participants]
  Yes | 24 | 28 | 52
  No | 7 | 8 | 15
On oral agents [Number; unit: participants]
  Yes | 20 | 24 | 44
  No | 11 | 12 | 23
On insulin [Number; unit: participants]
  Yes | 10 | 5 | 15
  No | 21 | 31 | 52
On other diabetes medications [Number; unit: participants]
  Yes | 2 | 3 | 5
  No | 29 | 33 | 62
Used diabetic supplies [Number; unit: participants]
  Yes | 18 | 10 | 28
  No | 13 | 26 | 39
Years since diabetes diagnosis [Mean (Standard Deviation); unit: years] | 8.0 (7.4) | 9.9 (10.3) | 9.0 (9.1)

OUTCOME MEASURES:

1. Primary Outcome: Change in Hemoglobin A-1C From Baseline
Description: Compare changes in Hemoglobin A-1C from baseline between the two groups.
Time Frame: baseline and 12 months
Population: Specific employers were recruited and offered waiver of out-of-pocket costs for diabetes-related care to their employees to participate in the study. The number of participants reported reflects only those participants who had both baseline and 12-month lab tests.
Measure: Mean (Standard Deviation); unit: percentage of glycolsylated hemoglobin
Groups:
- Pharmacists Consults Plus Out-of-pocket Cost Waiver: Employees received the same waiver of out-of-pocket expenses and also received up to 12 monthly visits with a pharmacist for consulting on monitoring and other educational aspects of diabetes self-management.
Arm/Group | Usual Care Plus Out-of-pocket Cost Waiver | Pharmacists Consults Plus Out-of-pocket Cost Waiver
Number analyzed (Participants) | 29 | 36
percentage of glycolsylated hemoglobin | -0.16 (0.42) | -0.50 (0.50)
Statistical Analysis 1: Comparison: Usual Care Plus Out-of-pocket Cost Waiver vs Pharmacists Consults Plus Out-of-pocket Cost Waiver; Null hypothesis is mean change in usual care group equals mean change in Empower group. Power calculation required 150 per group assuming 25% would withdraw prior to 12 months; Test type: Superiority or Other; p = 0.0757, ANCOVA — Adjusted for baseline Hemoglobin A-1C

2. Secondary Outcome: Changes From Baseline in LDL, HDL, Total Cholesterol, Triglycerides
Description: Changes from baseline in LDL, HDL, total cholesterol, triglycerides.
  Sample sizes for each individual test (usual care plus out-of-pocket cost waiver; EMPOWER group):
  1. LDL
  2. HDL
  3. Total cholesterol
  4. Triglycerides
Time Frame: baseline and 12 months
Population: The number of participants reported reflects only those participants who had both baseline and 12-month lab tests.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Usual Care Plus Out-of-pocket Cost Waiver | EMPOWER Group
Number analyzed (Participants) | 31 | 36
mg/dl
  LDL (n: 27; 35) | 0.1 [-8.3 to 8.5] | -3.9 [-17.0 to 9.2]
  HDL (n: 29; 36) | -3.6 [-7.2 to -0.05] | -6.3 [-9.1 to -3.4]
  Total cholesterol (n: 29; 36) | -5.1 [-16.5 to 6.3] | -11.6 [-25.0 to 1.8]
  triglycerides (n: 29; 36) | -5.8 [-58.3 to 46.6] | -8.9 [-30.0 to 12.3]
Statistical Analysis 1: Comparison: Usual Care Plus Out-of-pocket Cost Waiver vs EMPOWER Group; Comparison of change in LDL from baseline to 12 months between groups; Test type: Superiority or Other; p = 0.44, ANCOVA
Statistical Analysis 2: Comparison: Usual Care Plus Out-of-pocket Cost Waiver vs EMPOWER Group; Comparison of change in HDL from baseline to 12 months between groups; Test type: Superiority or Other; p = 0.16, ANCOVA
Statistical Analysis 3: Comparison: Usual Care Plus Out-of-pocket Cost Waiver vs EMPOWER Group; Comparison of change in total cholesterol from baseline to 12 months between groups; Test type: Superiority or Other; p = 0.14, ANCOVA
Statistical Analysis 4: Comparison: Usual Care Plus Out-of-pocket Cost Waiver vs EMPOWER Group; Comparison of change in triglycerides from baseline to 12 months between groups; Test type: Superiority or Other; p = 0.92, ANCOVA

3. Secondary Outcome: Changes in Economic Outcomes (Total Cost of Care, Cost of Diabetes Medications, Cost of Diabetes Supplies) From Baseline to 12 Months
Description: Changes in claims-based economic data on costs of total health care, diabetes medications, and diabetes supplies from baseline to 12 months. Only participants who had a claim in the 12 months prior to baseline were included in these analyses. The resulting sample sizes (usual care plus out-of-pocket cost waiver; EMPOWER group) for these outcomes are:
  1. Total cost of care
  2. Costs of diabetes medications
  3. Costs of diabetes supplies
Time Frame: baseline to 12 months
Population: Changes in claims-based data from baseline to 12 months among patients with at least one diabetes-related claim at baseline.
Measure: Mean (95% Confidence Interval); unit: US dollars
Arm/Group | Usual Care Plus Out-of-pocket Cost Waiver | Pharmacists Consults Plus Out-of-pocket Cost Waiver
Number analyzed (Participants) | 31 | 36
US dollars
  Total health care costs (n: 31; 36) | -89 [-3355 to 3177] | 1612 [-953 to 24176]
  Diabetes medication costs (n: 24; 28) | 516 [176 to 857] | 450 [69 to 830]
  Diabetes supplies costs (n: 18; 10) | 237 [59 to 415] | 191 [78 to 304]
Statistical Analysis 1: Comparison: Usual Care Plus Out-of-pocket Cost Waiver vs Pharmacists Consults Plus Out-of-pocket Cost Waiver; Comparison of change in cost of total health care from baseline to 12 months between groups. Analyses not adjusted for other variables; Test type: Superiority or Other; p = .3856, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Usual Care Plus Out-of-pocket Cost Waiver vs Pharmacists Consults Plus Out-of-pocket Cost Waiver; Comparison of change in cost of diabetes medications from baseline to 12 months between groups. Analyses not adjusted for other variables; Test type: Superiority or Other; p = .6413, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Usual Care Plus Out-of-pocket Cost Waiver vs Pharmacists Consults Plus Out-of-pocket Cost Waiver; Analyses not adjusted for other variables; Test type: Superiority or Other; p = .4303, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Change in Diabetes Knowledge and Empowerment (Patient Self-efficacy) From Baseline to 12 Months
Description: Psycho-social aspects of diabetes knowledge and empowerment. Sample sizes are in parentheses (usual care plus out-of-pocket cost waiver; EMPOWER group):
  1. Changes from baseline to 12 months for the Diabetes Empowerment Scale (DES). Mean score for 28 items each scored as a Likert scale from 1 to 5. Higher scores correspond to greater empowerment
  2. Changes from baseline to 12 months for the Adherence Starts with Knowledge (ASK-20) adherence barrier test total barrier score (TBC). The TBC has a range from 0 to 18 and higher scores correspond to greater barriers.
  3. Changes from baseline to 12 months for understanding of diabetes. This is a single question: "How would you rate your understanding of diabetes and its treatment?" which uses a 7-point scale Likert scale as the response from 1 (poor) to 7 (excellent).
Time Frame: From baseline to 12 months
Population: The number of participants reported for each outcome reflects those participants who completed both baseline and 12-month surveys.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Usual Care Plus Out-of-pocket Cost Waiver | EMPOWER
Number analyzed (Participants) | 31 | 36
units on a scale
  Overall Diabetes Empowerment Scale (n: 27; 34) | 0.29 [0.01 to 0.56] | 0.17 [0.04 to 0.30]
  Adherence Starts with Knowledge (ASK-20)(n:28; 31) | 0.25 [-0.76 to 1.26] | -0.65 [-1.86 to 0.57]
  Understanding of Diabetes (n: 29; 35) | -0.14 [-0.40 to 0.13] | 0.54 [0.12 to 0.96]
Statistical Analysis 1: Comparison: Usual Care Plus Out-of-pocket Cost Waiver vs EMPOWER; Comparison of change in Diabetes Empowerment Scale from baseline to 12 months between groups; Test type: Superiority or Other; p = 0.785, ANCOVA
Statistical Analysis 2: Comparison: Usual Care Plus Out-of-pocket Cost Waiver vs EMPOWER; Comparison of change in Adherence Starts with Knowledge (ASK-20) from baseline to 12 months between groups; Test type: Superiority or Other; p = 0.302, ANCOVA
Statistical Analysis 3: Comparison: Usual Care Plus Out-of-pocket Cost Waiver vs EMPOWER; Comparison of change in Understanding of Diabetes from baseline to 12 months between groups; Test type: Superiority or Other; p = 0.0024, ANCOVA

ADVERSE EVENTS:
Time Frame: Follow-up of approximately one year post-randomization (about 400 days, on average)
Arm/Group | Usual Care Plus Out-of-pocket Cost Waiver | EMPOWER Group
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/36
Other Adverse Events (participants affected / at risk) | 0/31 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No